CLINICAL TRIAL: NCT04594733
Title: The Effect of Minocycline and N-acetylcysteine for the Treatment of Fibromyalgia: a Double-blind, Randomized, Crossover Pilot Study
Brief Title: The Effect of Minocycline and N-acetylcysteine for the Treatment of Fibromyalgia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Michael Gabriel Hillegass, Associate Professor, Medical University of South Carolina
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 00102425
Record Dates: First submitted 2020-10-14; First posted 2020-10-20 (Actual); Results first posted 2024-01-30 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Fibromyalgia
MeSH Terms: conditions — Fibromyalgia | interventions — Minocycline

STUDY DESIGN:
Intervention Model Description: • A simple randomization method will be used to assign the initial treatment and then the opposite treatment will ensure for the second treatment period. Patients will be randomized to (i) 8 weeks of placebo, minimum 2 week washout period, and then 8 weeks of a combination minocycline (200 mg daily) and NAC (1200 mg daily) followed by a final 2 week washout or (ii) 8 weeks of a combination minocycline (200 mg daily) and NAC (1200 mg daily), minimum 2 week washout period, and then 8 weeks of placebo followed by a final 2 week washout.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo followed by minocycline (200 mg daily) and NAC (1200 mg daily) (Active Comparator): Participants will be randomized to 8 weeks of placebo, minimum 2 week washout period, and then 8 weeks of a combination minocycline (200 mg daily) and NAC (1200 mg daily) followed by a final 2 week washout
  Interventions: Drug: Placebo followed by minocycline (200 mg daily) and NAC (1200 mg daily)
- minocycline (200 mg daily) and NAC (1200 mg daily) followed by placebo (Active Comparator): Participants will be randomized to 8 weeks of a combination minocycline (200 mg daily) and NAC (1200 mg daily), minimum 2 week washout period, and then 8 weeks of placebo followed by a final 2 week washout
  Interventions: Drug: minocycline (200 mg daily) and NAC (1200 mg daily) followed by placebo

INTERVENTIONS:
Drug: minocycline (200 mg daily) and NAC (1200 mg daily) followed by placebo — minocycline (200 mg daily) and NAC (1200 mg daily) followed by placebo
  Arms: minocycline (200 mg daily) and NAC (1200 mg daily) followed by placebo
Drug: Placebo followed by minocycline (200 mg daily) and NAC (1200 mg daily) — Placebo followed by minocycline (200 mg daily) and NAC (1200 mg daily)
  Arms: Placebo followed by minocycline (200 mg daily) and NAC (1200 mg daily)

SUMMARY:
Evaluation of the effect of combinatorial treatment of fibromyalgia patients (standard of care + minocycline + N-acetylcysteine (NAC) relative to standard of care on subjective pain measurement Revised Fibromyalgia Impact Questionnaire (FIQR).

ELIGIBILITY:
Inclusion Criteria

* Female
* Age 18 years or older
* Diagnosis of fibromyalgia for at least 6 months (confirmed by the modified 2010 ACR Diagnostic Criteria for Fibromyalgia Widespread Pain Inventory and Symptom Severity Scale)
* Currently on birth control or unable to become pregnant
* Willingness to avoid taking opioid and opiate medications during the duration of the study (5-6 months) Exclusion Criteria
* Known hypersensitivity to minocycline or tetracycline antibiotics or to N-acetylcysteine
* Current opioid therapy or planned initiation of opioid therapy
* Active pregnancy, lactation or plans to become pregnant in the next 6 months
* Significant hepatic disease as indicated by an AST or ALT greater than twice the upper limits of normal or bilirubin greater than twice the upper limits of normal
* Significant renal disease as indicated by an estimated glomerular filtration rate less than 60 mL/min/1.73m2 at baseline or during the first washout period
* History of autoimmune syndromes (systemic lupus erythematosus, myasthenia gravis, rheumatoid arthritis,
* History of intracranial hypertension or pseudotumor cerebri
* History of IBD (Crohns disease, ulcerative colitis), Clostridium difficile infection
* History of esophagitis, esophageal obstruction, achalasia or esophageal dysmotility
* History of GI hemorrhage or known risk factors for GI hemorrhage, such as esophageal varices, peptic ulcer disease, etc.
* Subjects taking divalent and trivalent cations such as oral iron supplements, certain dietary supplements (multivitamins) that contain manganese or zinc, or antacids that contain aluminum, calcium, or magnesium, which would decrease minocycline absorption
* Subjects taking anticoagulant medication since minocycline can decrease plasma prothrombin activity
* Subjects taking isotretinoin
* Subject taking ergot alkaloids for migraines
* Subjects taking penicillin antibiotics
* Subjects taking methoxyflurane containing products
* Subjects who work outdoors or otherwise have prolonged exposure to UV light and sunlight
* Lack of access to reliable technology to be able to complete emailed REDCap questionnaires
* Cognitive deficits that may make it difficult to adhere to the medication regimen or provide consistent and timely completion of questionnaires
* Inability or unwillingness to give informed consent
* Unwillingness to use two forms of birth control for the entire duration of participation in the study (if capable of becoming pregnant)
* Unwillingness to complete home pregnancy tests throughout the study (if capable of becoming pregnant)
* Inability to swallow large pills

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2021-12-06 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael G Hillegass, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: First Intervention (8 Weeks)
Arm/Group | Placebo Followed by Minocycline (200 mg Daily) and NAC (1200 mg Daily) | Minocycline (200 mg Daily) and NAC (1200 mg Daily) Followed by Placebo
Started | 7 | 7
Received Intervention | 7 | 7
Completed | 7 | 3
Not Completed | 0 | 4
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Lost to Follow-up | 0 | 3
Period: First Washout (2 Weeks)
Arm/Group | Placebo Followed by Minocycline (200 mg Daily) and NAC (1200 mg Daily) | Minocycline (200 mg Daily) and NAC (1200 mg Daily) Followed by Placebo
Started | 7 | 3
Completed | 7 | 3
Not Completed | 0 | 0
Period: Second Intervention (8 Weeks)
Arm/Group | Placebo Followed by Minocycline (200 mg Daily) and NAC (1200 mg Daily) | Minocycline (200 mg Daily) and NAC (1200 mg Daily) Followed by Placebo
Started | 7 | 3
Completed | 5 | 3
Not Completed | 2 | 0
Not completed — Lost to Follow-up | 2 | 0
Period: Second Washout (2 Weeks)
Arm/Group | Placebo Followed by Minocycline (200 mg Daily) and NAC (1200 mg Daily) | Minocycline (200 mg Daily) and NAC (1200 mg Daily) Followed by Placebo
Started | 5 | 3
Completed | 5 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Followed by Minocycline (200 mg Daily) and NAC (1200 mg Daily) | Minocycline (200 mg Daily) and NAC (1200 mg Daily) Followed by Placebo | Total
Number analyzed (Participants) | 7 | 7 | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.3 (17.2) | 51.6 (9.98) | 48.4 (13.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 14
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 4 | 5 | 9
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Duration of Formal Diagnosis [Number; unit: participants]
  0-1 years | 0 | 2 | 2
  1-2 years | 1 | 1 | 2
  3-5 years | 1 | 0 | 1
  5-10 years | 4 | 3 | 7
  >10 years | 1 | 1 | 2
Duration of Symptoms [Number; unit: participants]
  1-2 years | 1 | 0 | 1
  3-5 years | 1 | 0 | 1
  5-10 years | 1 | 2 | 3
  >10 years | 4 | 5 | 9
Fibromyalgia Impact Questionnaire (FIQR) Score [Mean (Standard Deviation); unit: units on a scale] — The FIQR (Revised Fibromyalgia Impact Questionnaire) is comprised of 21 questions; 3 domains = function, overall impact, symptoms; 11-point numeric rating scale; questions framed with the context of the past 7 days. The instructions ask the patient to rate the difficulty on a scale of 0-10 (0 = No difficulty, and 10 = Very difficult) which indicates how much difficulty they have experienced in doing this activity during the past 7 days. The total FIQR score is the sum of each section. Range of scores are from 0-100. A lower score means a better outcome.
  units on a scale | 67.6 (12.9) | 58.4 (16.2) | 63.0 (14.9)
The Pain, Enjoyment of Life and General Activity (PEG) Score [Mean (Standard Deviation); unit: units on a scale] — In the PEG score, a higher score indicates more severe pain and pain-related interference. The PEG has 3 separate numerical scales. Each has ratings 0-10.The 1st scale asks individuals to rate their pain on average over the past week, the 2nd asks to rate how pain has interfered with their enjoyment of life in the past week, the 3rd asks to rate how pain has interfered with general activities. The total PEG scale is scored by adding each score and dividing by 3. The final score helps to track and monitor pain levels over time. The PEG score should decrease when treatment is effective.
  units on a scale | 7.29 (1.20) | 6.90 (1.74) | 7.10 (1.41)
Patient Health Questionnaire-2 (PHQ-2) Score [Median (Full Range); unit: units on a scale] — The PHQ-2 inquires about the frequency of depressed mood and anhedonia over the past two weeks. A PHQ-2 score ranges from 0-6. If the score is 3 or greater, major depressive disorder is likely.
  units on a scale | 4 [0 to 5] | 2 [0 to 5] | 2 [0 to 5]
Generalized Anxiety Disorder 2 (GAD-2) Score [Median (Full Range); unit: units on a scale] — The Generalized Anxiety Disorder 2-item (GAD-2) screens for generalized anxiety disorder 1. Two questions are asked, with the scoring of each ranging from 0-3, then both numbers added together. A total score of at least 3 points indicates possible anxiety disorder.
  units on a scale | 2 [0 to 6] | 2 [0 to 6] | 2 [0 to 6]
Widespread Pain Index (WPI) Score [Mean (Standard Deviation); unit: units on a scale] — The Widespread Pain Index (WPI) is a 19-point checklist that assesses pain or tenderness in 19 specific areas of the body within the past 7 days. Each area with pain receives point. The range in scores vary from 0-19, with 0 meaning no pain, and 19 meaning more areas of pain.
  units on a scale | 14.3 (3.90) | 10.6 (4.12) | 12.4 (4.31)
Symptom Severity Score (SS score) - Part 2a [Median (Full Range); unit: units on a scale] — Symptom Severity Score (SS Score) Part 2a assess symptom severity in the past 7 days in 3 categories, Fatigue, Waking unrefreshed, and cognitive symptoms. They are rated from 0 (no problem) to 3 (severe). Scores for each question are added up and used in part with section Symptom Severity 2b to get the total Symptom Severity Score. A lower score means less severe symptoms.
  units on a scale | 7 [6 to 9] | 5 [3 to 8] | 6 [3 to 9]
Symptom Severity (SS) 2b Score [Median (Inter-Quartile Range); unit: units on a scale] — Symptom Severity Score (SS Score) Part 2b asks individuals to check a box indicating if they have had any additional symptoms over the past week. The list of symptoms include items that are possible signs of fibromyalgia. The number of symptoms checked are scored as 1 point per check. If 0 symptoms = score of 0; 1 to 10 symptoms, = score of 1; 11 to 24 = score of 2; 25 or more symptoms = score of 3. A lower score means fewer symptoms.
  units on a scale | 1 [1 to 2] | 2 [1 to 2] | 1.5 [1 to 2]
Total Symptom Severity (SS) Score [Mean (Standard Deviation); unit: units on a scale] — Total Symptom Severity Score is derived using the score from Symptom Severity Score Part 2a, added to the score from Symptom Severity Score Part 2b. The Total SS ranges from 0-12, with 0 being little to no symptoms.
  units on a scale | 8.57 (1.9) | 7.14 (2.34) | 7.86 (2.18)

OUTCOME MEASURES:

1. Primary Outcome: Change in Revised Fibromyalgia Impact Questionnaire (FIQR) Score From Baseline to After Treatment Occurring at Weeks 8 and 18
Description: The FIQR (Revised Fibromyalgia Impact Questionnaire) is comprised of 21 questions spread across 3 domains: function, overall impact, symptoms, scored on an 11-point numeric rating scale. The questions are framed with the context of the past 7 days. The instructions ask the patient to rate the difficulty on a scale of 0-10 (0 = No difficulty, and 10 = Very difficult) which indicates how much difficulty they have experienced in doing the specified activity during the past 7 days. Each item is rated on a scale from 0 - 10, and the raw scores on each subscale. Then, the score on the function subscale is divided by 3, the overall impact subscale divided by 1, and the symptoms subscale divided by 2. These final scores from each subscale are then added up for the total FIQR score The total score can range from 0 -100. The total FIQR score is the sum of each section. A lower score means a better outcome. Higher scores indicate more severe impact.
Time Frame: Evaluated at baseline (prior to intervention) then again after treatment which occurs at week 8 and week 18
Measure: Mean (95% Confidence Interval); unit: Score
Groups:
- Placebo Treatment Period: Participants will be randomized to 8 weeks of placebo
- Minocycline (200 mg Daily) and NAC (1200 mg Daily) Treatment Period: Participants will be randomized to 8 weeks of a combination minocycline (200 mg daily) and NAC (1200 mg daily).
Arm/Group | Placebo Treatment Period | Minocycline (200 mg Daily) and NAC (1200 mg Daily) Treatment Period
Number analyzed (Participants) | 10 | 7
Score | 4.37 [-2.31 to 11.1] | 12.1 [6.30 to 17.9]

2. Secondary Outcome: Change in Pain, Enjoyment of Life and General Activity (PEG) Scale From Baseline to After Treatment Occurring at Weeks 8 and 18
Description: In the PEG score, a higher score indicates more severe pain and pain-related interference. The PEG has 3 separate numerical scales. Each has ratings 0-10.The first scale asks individuals to rate their pain, on average, over the past week, the second asks to rate how pain has interfered with their enjoyment of life in the past week, the third asks individuals to rate how pain has interfered with general activities. The PEG scale is scored by averaging the three numbers. The final score helps to track and monitor pain levels over time. The PEG score should decrease when treatment is effective.
Time Frame: Evaluated at baseline (prior to intervention) then again after treatment which occurs at week 8 and week 18
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Placebo Treatment Period | Minocycline (200 mg Daily) and NAC (1200 mg Daily) Treatment Period
Number analyzed (Participants) | 10 | 7
score on a scale | 0.64 [-0.36 to 1.64] | 1.24 [0.37 to 2.12]

3. Secondary Outcome: Change in Patient Health Questionnaire (PHQ-2) From Baseline to After Treatment Occurring at Weeks 8 and 18
Description: The change in depression scale (PHQ-2) by evaluating the number of days the participant feels down, depressed or hopeless and has little interest or pleasure in doing things rated as not at all (0), several days (1), more than half the days (2), or nearly every day (3) by scoring the 2 questions from 0-3 as indicated. Scores range from 0-6, with the higher score meaning the patient experiencing more severe symptoms.
Time Frame: Evaluated at baseline (prior to intervention) then again after treatment which occurs at week 8 and week 18
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Placebo Treatment Period | Minocycline (200 mg Daily) and NAC (1200 mg Daily) Treatment Period
Number analyzed (Participants) | 10 | 7
score on a scale | 0.12 [-0.55 to 0.80] | 0.23 [-0.38 to 0.84]

4. Secondary Outcome: Change in General Anxiety Disorder (GAD-2) Score From Baseline to After Treatment Occurring at Weeks 8 and 18
Description: The Generalized Anxiety Disorder 2-item (GAD-2) screens for generalized anxiety disorder 1. Two questions are asked, with the scoring of each ranging from 0-3, then both numbers added together, with possible scores ranging from 0-6. A total score of at least 3 points indicates possible anxiety disorder. The higher the score, the more severe anxiety.
Time Frame: Evaluated at baseline (prior to intervention) then again after treatment which occurs at week 8 and week 18
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Placebo Treatment Period | Minocycline (200 mg Daily) and NAC (1200 mg Daily) Treatment Period
Number analyzed (Participants) | 10 | 7
score on a scale | -0.02 [-0.70 to 0.66] | 0.72 [0.10 to 1.33]

5. Secondary Outcome: Patient Global Impression of Change (PGIC)
Description: Patient Global Impression of Change (PGIC) has the subject will reporting whether there was a change in their activity, limitations, symptoms, emotions and overall quality of life by rating "no change", "almost the same", "a little better", "somewhat better", "moderately better", "better" or "a great deal better". Participants will also rate degrees of change from much better (0), 5 (no change), to much worse (10). The higher the score, the worse their impression of their health status was worse than previously. Scores will range from no change to a great deal better, and from 0 (much better) to 10 (much worse).
Time Frame: immediately after each treatment at week 8 (first intervention) and week 18 (second intervention)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo Treatment Period | Minocycline (200 mg Daily) and NAC (1200 mg Daily) Treatment Period
Number analyzed (Participants) | 10 | 7
units on a scale | 1.6 (0.72) | 2.8 (0.79)

6. Other Pre Specified Outcome: Modified 2010 American College of Rheumatology Preliminary Diagnostic Criteria for Fibromyalgia (Modified ACR 2010)
Description: Participants will rate change using modified 2010 American College of Rheumatology Preliminary Diagnostic Criteria for Fibromyalgia (modified ACR 2010) by answering questions related to their areas of pain, amount of medication required for pain, and symptoms.
Time Frame: Evaluated at baseline (prior to intervention) then again after treatment which occurs at week 8 and week 18
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse event data was collected weekly from weeks 1-19.
Groups:
- Placebo: Participants will be randomized to 8 weeks of placebo, minimum 2 week washout period, and then 8 weeks of a combination minocycline (200 mg daily) and NAC (1200 mg daily) followed by a final 2 week washout
  Placebo followed by minocycline (200 mg daily) and NAC (1200 mg daily): Placebo followed by minocycline (200 mg daily) and NAC (1200 mg daily)
- Minocycline 200 mg Daily + NAC 1200mg Daily: Participants will be randomized to 8 weeks of a combination minocycline (200 mg daily) and NAC (1200 mg daily), minimum 2 week washout period, and then 8 weeks of placebo followed by a final 2 week washout
  minocycline (200 mg daily) and NAC (1200 mg daily) followed by placebo: minocycline (200 mg daily) and NAC (1200 mg daily) followed by placebo
Arm/Group | Placebo | Minocycline 200 mg Daily + NAC 1200mg Daily
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/14
Other Adverse Events (participants affected / at risk) | 5/10 | 8/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=10) | Minocycline 200 mg Daily + NAC 1200mg Daily (N=14)
Malaise (General disorders) | 1 (1) | 5 (5)
Other (General disorders) | 2 (2) | 1 (1) — Other
Drowsiness (General disorders) | 0 (0) | 3 (3)
Light headedness (Nervous system disorders) | 1 (1) | 2 (2)
Vertigo (Nervous system disorders) | 1 (1) | 1 (1)
Photosensitivity (Nervous system disorders) | 1 (1) | 2 (2)
Pain with swallowing (Gastrointestinal disorders) | 1 (1) | 0 (0)
Muscle Pain (General disorders) | 2 (2) | 4 (4)
Joint Pain (General disorders) | 1 (1) | 5 (5)
Joint Swelling (General disorders) | 1 (1) | 2 (2)
Fatigue (General disorders) | 1 (1) | 3 (3)
Red Itchy Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dizziness (General disorders) | 0 (0) | 3 (3)
Ear Ringing (General disorders) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 1 (1) | 3 (3)
Blurry Vision (Nervous system disorders) | 0 (0) | 2 (2)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (General disorders) | 0 (0) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Itchiness (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Facial Flushing (General disorders) | 0 (0) | 1 (1)
Sun Burn (General disorders) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-12-02): https://cdn.clinicaltrials.gov/large-docs/33/NCT04594733/Prot_SAP_000.pdf